CLINICAL TRIAL: NCT00245843
Title: Vermont Intervention: Effect on Joint Attention Skills Between Parents and Moderate/Late Preterm Infants Int the First Year of Life
Brief Title: Vermont Intervention: Effect on Joint Attention Skills Between Parents and Moderate/Late Preterm Infants in the First Year of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ullevaal University Hospital (Other)
Collaborators: The Royal Norwegian Ministry of Health (Other); Regionsenter for barn og unges psykiske helse (Other); Norwegian Nurses Association (NSF) (Unknown); University of Oslo (Other)
Responsible Party: South-Eastern Norway Regional Health Authority, South-Eastern Norway Regional Health authority
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Vermont
Record Dates: First submitted 2005-10-27; First posted 2005-10-28 (Estimated); Last update posted 2009-04-01 (Estimated); Status verified 2009-03

CONDITIONS: Premature Birth
Keywords: Premature birth; moderate preterm; late preterm; Joint attention; Social interaction; Child development; Parent; infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Mother Infant Transaction Program (MITP) — Psychosocial intervention. 11-session one hour standardized intervention program. The aim of the MITP is to help parents to appreciate their infant's unique characteristics,temperament and developmental potential.

SUMMARY:
The purpose of this study is to investigate if the effects of the Vermont intervention, implemented by nurses in a Neonatal Intensive Care Unit (NICU), can influence social interaction and joint attention skills between parents and preterm babies in the second half of the first year of life.

DETAILED DESCRIPTION:
The bases of parental sensitivity and infants' joint attention skills are probably established during the child's first year of life. Research suggests that the quality of early social interaction is related to children's later development and mental health. Preterm infants are at risk for developing interaction disturbances in the first year of life, and such aberrancies often lay the foundation for later problems of adaptation. Following preterm birth the infant is exposed to an atypical extra uterine environment. In such an environment it is hard for an immature brain to modulate the infant's behaviour properly.

Under such circumstances there are several factors to consider. The disturbances that may be seen later may be mediated and moderated by the infant's state, parental circumstances and conditions in the hospital environment. Parents of preterm infants experience interruption of normal pregnancy and may be in a difficult emotional state after preterm birth, and often they are not prepared for their role as parents. They are also vulnerable to stress and worries concerning survival of their baby. These conditions are assumed to have a negative influence on the social interaction between preterm infant and parents, and can make it difficult for the caretakers to adapt to their low birth weight infant and to engage in social interaction with their baby.

The purpose of this study is to evaluate the effects of a neonatal intervention program (Vermont-intervention) on parental sensitivity and the interaction skills between parents and preterm babies in the first year of life. The intervention is based on a transactional model of development, which emphasizes the mutual regulation and interaction going on between a child and its caretakers over time.

The study is a randomized controlled trial in a NICU environment. 100 preterm children born between 30 and 36 weeks of gestation are randomly assigned to a control group and an experimental group. The intervention is the Mother Infant Transaction Program (MITP) called the Vermont intervention. In addition, 50 full term normal-weight infants are recruited into a full term control group. The work of recruitment and randomizing of the 150 families to the three groups is carried out by a paediatric research assistant who will also be responsible for the organization and implementation of the interventions at hospital and at home after discharge from hospital. To the extent it is possible, the nurse researcher is not supposed to recognize the group identity of the participants in the three groups when administering questionnaires and scoring video recordings of social interaction and joint attention between mother and child at ages 6, 9 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Preterm newborns with gestational age > 29.6 and < 36.0 weeks at birth.
* Full term newborns with gestational age > 36.9 weeks at birth and birth weight equal to or more than 2500 grams
* Admitted to Ullevål University Hospital
* Families are recruited to the study before infants are discharged from the hospital

Exclusion Criteria:

* Congenital or chromosomal abnormality, and/or severe neonatal diseases
* History of maternal substance or psychiatric disorders.

Min Age: 30 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2005-01; Primary Completion 2008-02 (Actual); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Social interaction and joint attention skills between parents and moderate/late preterm infants within first year of life | 1, 4, 6, 9 and 12 months
Child outcome: child's quality and social capacity for joint attention/social interaction | 1,4, 9 and 12 months
Parenting outcome: parents' sensitivity/responsitivity to children's behaviour/signals, parental stress | 1, 4, 6, 9 and 12 months

SECONDARY OUTCOMES:
Child outcomes: child development, child temperament, growth | 1, 4, 6, 9 and 12 months
Parenting outcome: depression, stress, maternal confidence | 1, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Lindemann, MD, PhD, Study Director — Ullevål University Hospital (UUS)
Locations (1):
- Ullevaal University Hospital (UUS), Oslo, Norway

REFERENCES:
- [Derived] Ravn IH, Smith L, Smeby NA, Kynoe NM, Sandvik L, Bunch EH, Lindemann R. Effects of early mother-infant intervention on outcomes in mothers and moderately and late preterm infants at age 1 year: a randomized controlled trial. Infant Behav Dev. 2012 Feb;35(1):36-47. doi: 10.1016/j.infbeh.2011.09.006. Epub 2011 Oct 22. PMID 22024475
- [Derived] Ravn IH, Smith L, Lindemann R, Smeby NA, Kyno NM, Bunch EH, Sandvik L. Effect of early intervention on social interaction between mothers and preterm infants at 12 months of age: a randomized controlled trial. Infant Behav Dev. 2011 Apr;34(2):215-25. doi: 10.1016/j.infbeh.2010.11.004. Epub 2011 Mar 2. PMID 21371754